CLINICAL TRIAL: NCT02050360
Title: Efficacy and Safety of "as Required" Sildenafil for Patients With Moderate to Severe Raynaud's Phenomenon (RP)
Brief Title: "As Required" Oral Sildenafil in Raynaud's Phenomenon
Acronym: PROFIL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCIC/12/26; 2013-000014-38 (EudraCT Number); 12G01 (Other: Promotor)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Raynaud's Phenomenon
Keywords: Raynaud's phenomenon; Sildenafil; Systemic Sclerosis; Local cooling; Microcirculation
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Systemic | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sildenafil 80 mg (Experimental): Sildenafil 80 mg
  Interventions: Drug: Sildenafil 80 mg
- Sildenafil 40 mg (Experimental): Sildenafil 40 mg
  Interventions: Drug: Sildenafil 40 mg
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil 40 mg
  Arms: Sildenafil 40 mg
Drug: Sildenafil 80 mg
  Arms: Sildenafil 80 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether "on-demand" sildenafil is effective in the treatment of Raynaud's phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Active Raynaud's Phenomenon characterized by a clinical history of primary or secondary Raynaud's Phenomenon
* At least 7 RP attacks per week on 5 or more days per week (assessed over the 2 weeks preceding inclusion)
* Patients who have dated and signed the informed consent form
* Contraception for women

Exclusion Criteria:

* Recently diagnosed RP (less than 2 months).
* Uncontrolled hypertension, diabetes mellitus, angina
* Haemodynamic instability
* Nonarteritic ischemic optic neuropathy
* Pulmonary hypertension
* Subjects currently taking sildenafil, tadalafil or vardenafil
* Subjects currently taking nitrates
* Subjects currently taking strong CYP3A inhibitors
* Pregnancy (or considering pregnancy in the next 4 months)
* Breast feeding
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Mean change in the Raynaud's Condition Score (RCS) during treatment, as compared to placebo. | 7 days
  RCS is self-reported every day and averaged over 7-day periods

SECONDARY OUTCOMES:
Frequency of RP: number of RP attacks during treatment, as compared to placebo. | 7 days
  An attack is defined as an episode of pallor or cyanosis (with or without pain,tingling or numbness). The number of attacks is self-reported every day and averaged over 7-day periods
Patients' preference: comparison between the number of patients favoring a treatment to another. | Every 3 weeks of treatment (week 3, 6 and 9)
Pain associated with RP: Mean change in the Raynaud's pain score during treatment, as compared to placebo. | 7 days
  Pain associated with each attack is self-reported on a 10-point scale, and averaged over 7-day periods
Frequency and severity of adverse drug events during treatment, as compared to placebo | 7 days
Microvascular reactivity: index of skin perfusion in response to local/regional cooling after a single dose of sildenafil, as compared to placebo (laboratory experiments) | Week 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc CRACOWSKI, MD, Principal Investigator — INSERM CIC03 - Unité de Pharmacologie Clinique
Locations (1):
- Clinical Investigation Center - Pharmacology Unit - University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Derived] Maltez N, Maxwell LJ, Rirash F, Tanjong Ghogomu E, Harding SE, Tingey PC, Wells GA, Tugwell P, Pope J. Phosphodiesterase 5 inhibitors (PDE5i) for the treatment of Raynaud's phenomenon. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD014089. doi: 10.1002/14651858.CD014089. PMID 37929840
- [Derived] Roustit M, Giai J, Gaget O, Khouri C, Mouhib M, Lotito A, Blaise S, Seinturier C, Subtil F, Paris A, Cracowski C, Imbert B, Carpentier P, Vohra S, Cracowski JL. On-Demand Sildenafil as a Treatment for Raynaud Phenomenon: A Series of n-of-1 Trials. Ann Intern Med. 2018 Nov 20;169(10):694-703. doi: 10.7326/M18-0517. Epub 2018 Oct 30. PMID 30383134